CLINICAL TRIAL: NCT01876836
Title: Comparation the Effect of C-LMA and I-gel in Regurgitation and Postoperative Complications
Brief Title: Clasic Laryngeal Mask Airway(C-LMA) and I-gel Releated Regurgitation and Complications
Acronym: C-LMA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Reyhan Polat, Doctor, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single
Record Dates: First submitted 2013-06-10; First posted 2013-06-13 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Bladder Tumour; Prostate Hyperplasia
Keywords: i-gel; C-LMA; gastroeosephageal reflux; sore troat
MeSH Terms: conditions — Urinary Bladder Neoplasms; Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- i-gel (Experimental): i-gel placed after induction
  Interventions: Device: i-gel
- C-LMA (Active Comparator): C-LMA placed after induction
  Interventions: Device: C-LMA

INTERVENTIONS:
Device: i-gel — i-gel placed after induction
  Other Names: supraglottic airway device
  Arms: i-gel
Device: C-LMA — placed after induction
  Other Names: supraglottic airway device
  Arms: C-LMA

SUMMARY:
1. i-gel
2. C-LMA

Compare the effect on gastroeosephageal reflux Postoperative complicatios.

DETAILED DESCRIPTION:
120 ASA I-II adult patients. Patients were randomised into two groups

1. i-gel
2. C-LMA Volume controlled ventilation, general anesthesia Asses Gastroeosephageal reflux, sore throat, coughing, dysphagia,dysphonia recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Adult
* Elective surgery
* Bladder tumour
* Prostat hyperplasi

Exclusion Criteria:

* Emergency surgery
* Hiatal hernia
* Gastroeosephageal reflux disease

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-07; Primary Completion 2013-08 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Ph MEASUREMENT | 1 MİNUTE AFTER EXTUBATİON
  The ph of the secretions on the airway device will be measurd with a Ph-meter

SECONDARY OUTCOMES:
Bleu dye on the airway device | 5 min after placenent
  The airway device will be examined with fiberoptic endoscope after placement

OTHER OUTCOMES:
Blue dye on airway device | 1 min after extubation
  the airway device will be examined for a precence of blue dye

CONTACTS AND LOCATIONS:
Overall Officials: Reyhan Polat, MD, Principal Investigator — Diskapi Yildirim Beyazit Education and Research Hospital
Locations (1):
- DiskapiYBERH, Ankara, Altındağ, Turkey (Türkiye)